CLINICAL TRIAL: NCT04157478
Title: Addition of Anlotinib Hydrochloride to the Stupp Regimen Versus the Stupp Regimen Alone for Newly Diagnosed Glioblastoma: A Randomized Multicenter Prospective Phase II Study
Brief Title: Addition of Anlotinib Hydrochloride to the Stupp Regimen Versus the Stupp Regimen Alone for Newly Diagnosed Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Cancer Hospital of Guangxi Medical University (Other); Liuzhou Workers' Hospital (Other Government); Nanxishan Hospital (Unknown); LiuZhou People's Hospital (Other); Affiliated Hospital of Guilin University (Unknown)
Responsible Party: Principal Investigator, Heming Lu, Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GXPH-19001
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Anlotinib hydrochloride; Stupp regimen; Temozolomide; Radiation therapy; Tyrosine kinase inhibitor
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation therapy, Temozolomide and anlotinib (Experimental): Patients will receive standard radiation therapy plus temozolomide (Stupp regimen). Anlotinib hydrochloride will be given with a daily dose of 12 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Interventions: Drug: Anlotinib Hydrochloride; Radiation: Radiation therapy; Drug: Temozolomide
- Radiation therapy and temozolomide (Active Comparator): Patients will receive standard radiation therapy plus temozolomide (Stupp regimen).
  Interventions: Radiation: Radiation therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib hydrochloride will be given with a daily dose of 12 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Arms: Radiation therapy, Temozolomide and anlotinib
Radiation: Radiation therapy — Radiation therapy will be delivered in daily fractions of 2 Gy given 5 days a week for a total of 60 Gy.
Drug: Temozolomide — Temozolomide will be administered at a daily dose of 75 mg/m2 until the completion of radiation therapy. Four weeks after the completion of radiation therapy, patients will be given with adjuvant chemotherapy with temozolomide at a dose of 150-200 mg/m2 for 5 days of a 28-day cycle for a total of 6 cycles.

SUMMARY:
For patients with glioblastoma,postoperative radiotherapy combined with concurrent and adjuvant temozolomide (Stupp regimen) has long been considered a standard treatment approach.The treatment outcomes, however, are still dismal, with a median overall survival time of 8-12 months. As a novel small molecule multi-target tyrosine kinase inhibitor, anlotinib hydrochloride has been found to be able to inhibit both tumor angiogenesis and cell growth.Previous studies on recurrent glioblastoma have demonstrated its effectiveness in tumor control with manageable toxicities. The current study is designed to evaluate the efficacy and feasibility of the additional anlotinib hydrochloride to the Stupp regimen for newly diagnosed glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and histological proven glioblastoma
* Complete gross resection or subtotal resection
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate bone marrow, liver and renal function
* Written informed consent

Exclusion Criteria:

* Meningeal carcinomatosis or spinal compression
* Patients who have previously received chemotherapy, targeted therapy, or anti-angiogenesis
* Active, known, or suspected autoimmune disease
* Severe allergy to anlotinib or temozolomide
* Patient having acute hepatitis virus infection, active tuberculosis, or other acute infectious diseases
* Uncontrolled mental disorders
* High risk of bleeding
* Severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms), according to NYHA criteria; grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%
* Contraindicated for MRI examination
* Recipient of live vaccine prior to the first dose of anlotinib
* Ready for or previously received organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
Objective response rate | 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - Liuzhou Worker's Hospital, Liuchow, Guangxi
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Yulin First Hospital, Yulin, Guangxi